CLINICAL TRIAL: NCT00002536
Title: TREATMENT OF PATIENTS WITH SUBOPTIMAL ('BULKY') STAGE IB CARCINOMA OF THE CERVIX: A RANDOMIZED COMPARISON OF RADICAL HYSTERECTOMY AND PELVIC AND PARA-AORTIC LYMPHADENECTOMY WITH OR WITHOUT NEOADJUVANT VINCRISTINE AND CISPLATIN CHEMOTHERAPY, PHASE III
Brief Title: Surgery With or Without Chemotherapy in Treating Patients With Stage IB Cervical Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000078470; GOG-141
Record Dates: First submitted 1999-11-01; First posted 2004-03-26 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2008-03

CONDITIONS: Cervical Cancer
Keywords: stage IB cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Vincristine; Surgical Procedures, Operative; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: vincristine sulfate
Procedure: surgical procedure
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving chemotherapy drugs before surgery may shrink the tumor so that it can be removed during surgery.

PURPOSE: Randomized phase III trial to compare surgery with or without chemotherapy in treating patients who have stage IB cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare disease free survival, overall survival, and local control in patients with bulky stage IB carcinoma of the cervix treated with radical hysterectomy and pelvic and para-aortic lymphadenectomy with or without neoadjuvant vincristine and cisplatin. II. Compare adverse effects of radical hysterectomy and pelvic and para-aortic lymphadenectomy with or without neoadjuvant vincristine and cisplatin in these patients.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms. Arm I: Surgery. All patients undergo intra-abdominal and retroperitoneal exploratory laparotomy. Patients without metastases also undergo radical hysterectomy with pelvic and para-aortic lymphadenectomy. Beginning 2-4 weeks after surgery, patients with 1 or more positive lymph nodes or positive surgical margins on the radical hysterectomy specimen receive adjunctive radiotherapy 5 days each week for 4-6 weeks. Patients with histologically confirmed metastases do not undergo radical hysterectomy with pelvic and para-aortic lymphadenectomy, but receive radiotherapy 5 days each week for 6-8 weeks beginning 2-4 weeks after the laparotomy. Patients who undergo radiotherapy also receive cisplatin IV over 1 hour on days when radiotherapy is administered for up to 6 doses of cisplatin. Arm II: Patients receive vincristine IV bolus immediately followed by cisplatin IV over 1 hour on days 1, 11, and 21. Courses repeat every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Beginning approximately 4 weeks after the last doses of neoadjuvant vincristine and cisplatin, patients receive surgery, radiotherapy, and cisplatin as in Arm I. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 170-340 patients will be accrued for this study over approximately 4.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Previously untreated, histologically proven invasive carcinoma of the cervix Eligible histologies: Squamous Adenocarcinoma Adenosquamous Eligible stages: Bulky stage IB, i.e.: Exophytic lesions 4 cm or greater in diameter OR Cervix expanded to 4 cm or greater and presumed clinically to result from cancer No extension beyond cervix clinically and by IVP or CT with contrast

PATIENT CHARACTERISTICS: Age: Not specified Performance status: GOG 0-2 Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times normal AST no greater than 3 times normal Alkaline phosphatase no greater than 3 times normal Renal: Creatinine no greater than 2.0 mg/dL Other: No septicemia or severe infection No other concurrent malignancy within the past 5 years except curatively treated nonmelanomatous skin cancer and prior malignancy therapy does not contraindicate current protocol therapy Suitability for radical hysterectomy and lymphadenectomy required

PRIOR CONCURRENT THERAPY: No prior therapy for cervical cancer No prior pelvic irradiation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-12; Primary Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary L. Eddy, MD, Study Chair — Kaiser Permanente Medical Center - Bellflower
Locations (41):
- United States (41):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Southern California Permanante Medical Group, Bellflower, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Community Hospital of Los Gatos, Los Gatos, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Tufts University School of Medicine, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Brookview Research, Inc., Nashville, Tennessee
  - Fletcher Allen Health Care, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington

REFERENCES:
- [Result] Eddy GL, Bundy BN, Creasman WT, Spirtos NM, Mannel RS, Hannigan E, O'Connor D. Treatment of ("bulky") stage IB cervical cancer with or without neoadjuvant vincristine and cisplatin prior to radical hysterectomy and pelvic/para-aortic lymphadenectomy: a phase III trial of the gynecologic oncology group. Gynecol Oncol. 2007 Aug;106(2):362-9. doi: 10.1016/j.ygyno.2007.04.007. Epub 2007 May 9. PMID 17493669